CLINICAL TRIAL: NCT03390946
Title: Feasibility Study of Interval Compressed Regimen Using Four-drugs for Osteosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Byung-Kiu Park (Other Government)
Collaborators: Samsung Medical Center (Other); Chungnam National University Hospital (Other)
Responsible Party: Sponsor-Investigator, Byung-Kiu Park, Prof., National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-OSA-1601
Record Dates: First submitted 2017-12-11; First posted 2018-01-05 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Osteosarcoma; Feasibility; Treatment Response; Biomarker
Keywords: four-drugs, interval-compression
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- four-drug interval-compressed regimen (Experimental): Interventions for 'four-drug interval-compressed regimen': Drug: methotrexate, cisplatin, doxorubicin, ifosfamide.
  Newly diagnosed oseteosarcoma patients under 40 years are eligible. Neoadjuvant chemotherapy with four drugs in an interval-compressed schedule will be done as a single arm.
  Duration of neoadjuvant chemotherapy will be 10 weeks like that of conventional three-drug regimen, although four-drugs are employed in the current protocol.
  After tumor resection operation, participants will be divided to poor responder group and good responder group based on 90% necrosis rate of a tumor specimen.
  Poor responder group and will be assigned to 'Poor responder group adjuvant chemotherapy' and good responder will be assigned to 'Good responder group adjuvant chemotherapy'.
  Interventions: Drug: Poor responder group adjuvant chemotherapy; Drug: Good responder group adjuvant chemotherapy

INTERVENTIONS:
Drug: Poor responder group adjuvant chemotherapy — Poor responder group (necrosis ≤ 90%)
  : week 0, 7 and 14, doxorubicin; week 2, 9 and 16, ifosfamde, week 4, 11, 18 and 19, methotrexate; wk 5, 12 and 20
  B. Resection of tumor
  C. Adjuvant chemotherapy
  1. Poor responder group (necrosis ≤ 90%)
     * week 0, 7 and 14, doxorubicin; week 2, 9 and 16, ifosfamde, week 4, 11, 18 and 19, methotrexate; wk 5, 12 and 20
  2. Good responder group (necrosis > 90%)
     * week 0 and 8, doxorubicin; week 2 and 10, ifosfamide; week 4, 5, 12 and 13, methotrexate; week 6 and 14, cisplatin
  Other Names: PR adjuvant four-drug interval-compressed regimen
Drug: Good responder group adjuvant chemotherapy — Good responder group (necrosis > 90%)
  : week 0 and 8, doxorubicin; week 2 and 10, ifosfamide; week 4, 5, 12 and 13, methotrexate; week 6 and 14, cisplatin
  Other Names: GR adjuvant four-drug interval-compressed regimen

SUMMARY:
The aim of the study is to test the feasibility of four-drug, interval-compressed regimen in osteosarcoma.

Primary objective is to explore the toxicity and mortality related to treatment. Secondary objectives are to examine tumor necrosis rates after neoadjuvant chemotherapy, and to evaluate the usefulness of circulating cell-free DNA, survivin, or transforming growth factor-beta1 levels as well as programmed cell death ligand 1 expression in tumor specimen as a predictive or prognostic biomarker in osteosarcoma patients.

DETAILED DESCRIPTION:
In this study, the investigators will investigate the feasibility of interval compressed regimen using four-drugs in newly-diagnosed osteosarcoma patients. Four drugs will be adriamycin, high-dose methotrexate, cisplatin, ifosfamide. All these drugs will be given preoperatively in an interval-compressed schedule, but postoperatively at a regular interval. Neoadjuvant therapy will be composed of two courses, and adjuvant therapy of two or three courses depending on necrosis rates following neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed osteosarcoma patients under age 40 years.

Exclusion Criteria:

* Patients who don't meet the organ function criteria as follows;

  1. renal function : CCr or GFR or eGFR ≥ 70 mL/min/1.73 m2
  2. liver function : AST/ALT ≤ 5 x upper limit, total bilirubin ≤ 1.5 x upper limit of normal for age
  3. cardiac function : shortening fraction ≥ 24% or ejection fraction ≥ 50% (Echo)
  4. lung function : No dyspnea on rest, If dyspnea exists, SpO2 95% or more in room air by pulse oximetry,
  5. hematologic : ANC ≥ 750/uL and platelet ≥ 75,000/uL

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity determined according to CTCAE | Until study completion, an average of 3 years
  treatment-related toxicity (organ dysfunction, neutropenic fever, infection, mortality, et al.)

SECONDARY OUTCOMES:
tumor necrosis rate | Until study completion, an average of 3years
  necrosis rate of the excised tumor after neoadjuvant chemotherapy
Predictive or prognostic biomarker | Until study completion, an average of 3 years
  Usefulness of circulating cell-free DNA, survivin, transforming growth factor-beta1 levels and programmed cell death 1 expression in tumor specimen as a biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Kiu Park, M.D., Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Clinical data of individual participants can be shared without personal information. Each participating center will submit the clinical data to the principal investigation center, after eliminating personal data.

REFERENCES:
- [Background] Lewis IJ, Nooij MA, Whelan J, Sydes MR, Grimer R, Hogendoorn PC, Memon MA, Weeden S, Uscinska BM, van Glabbeke M, Kirkpatrick A, Hauben EI, Craft AW, Taminiau AH; MRC BO06 and EORTC 80931 collaborators; European Osteosarcoma Intergroup. Improvement in histologic response but not survival in osteosarcoma patients treated with intensified chemotherapy: a randomized phase III trial of the European Osteosarcoma Intergroup. J Natl Cancer Inst. 2007 Jan 17;99(2):112-28. doi: 10.1093/jnci/djk015. PMID 17227995
- [Background] Marina NM, Smeland S, Bielack SS, Bernstein M, Jovic G, Krailo MD, Hook JM, Arndt C, van den Berg H, Brennan B, Brichard B, Brown KLB, Butterfass-Bahloul T, Calaminus G, Daldrup-Link HE, Eriksson M, Gebhardt MC, Gelderblom H, Gerss J, Goldsby R, Goorin A, Gorlick R, Grier HE, Hale JP, Hall KS, Hardes J, Hawkins DS, Helmke K, Hogendoorn PCW, Isakoff MS, Janeway KA, Jurgens H, Kager L, Kuhne T, Lau CC, Leavey PJ, Lessnick SL, Mascarenhas L, Meyers PA, Mottl H, Nathrath M, Papai Z, Randall RL, Reichardt P, Renard M, Safwat AA, Schwartz CL, Stevens MCG, Strauss SJ, Teot L, Werner M, Sydes MR, Whelan JS. Comparison of MAPIE versus MAP in patients with a poor response to preoperative chemotherapy for newly diagnosed high-grade osteosarcoma (EURAMOS-1): an open-label, international, randomised controlled trial. Lancet Oncol. 2016 Oct;17(10):1396-1408. doi: 10.1016/S1470-2045(16)30214-5. Epub 2016 Aug 25. PMID 27569442